CLINICAL TRIAL: NCT02020512
Title: A Study of 0.03% Bimatoprost in the Treatment of Primary Open Angle Glaucoma and Ocular Hypertension
Acronym: LOTUSDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-BIM-1102
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.03% Bimatoprost (Experimental): 0.03% bimatoprost (LUMIGAN®) 1 drop in the affected eye once daily in the evening as monotherapy or adjunctive therapy for 5 weeks.
  Interventions: Drug: 0.03% Bimatoprost

INTERVENTIONS:
Drug: 0.03% Bimatoprost — 0.03% bimatoprost (LUMIGAN®) 1 drop in the affected eye once daily in the evening as monotherapy or adjunctive therapy for 5 weeks.
  Other Names: LUMIGAN®

SUMMARY:
This study will evaluate 0.03% bimatoprost in the treatment of primary open angle glaucoma and ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension
* No use of Lumigan® in the past 3 months

Exclusion Criteria:

* Received laser therapy, glaucoma surgery, cataract surgery, or other ocular surgery within the past 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Guangzhou, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.03% Bimatoprost
Started | 87
Completed | 79
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | 0.03% Bimatoprost
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.3 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase (worsening).
Time Frame: Baseline, Week 5
Population: Intent-to-Treat: all treated patients
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | 0.03% Bimatoprost
Number analyzed (Participants) | 87
Millimeters of Mercury (mmHg)
  Baseline | 22.2 (5.3)
  Change from Baseline at Week 5 | -6.7 (4.5)

ADVERSE EVENTS:
Arm/Group | 0.03% Bimatoprost
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 67/87
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.03% Bimatoprost (N=87)
Conjunctival Hyperemia (Eye disorders) | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.